CLINICAL TRIAL: NCT01366274
Title: Comparison of Protective Manual Hyperinflation With Current Methods in Ventilated Acute Trauma Patients: a Randomized Controlled Trial
Brief Title: Protective Manual Hyperinflation in Acute Mechanically Ventilated Trauma Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Queensland (Other)
Collaborators: Royal Brisbane and Women's Hospital (Other Government)
Responsible Party: Dr Jennifer Paratz, University of Queensland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PMH1
Record Dates: First submitted 2011-05-31; First posted 2011-06-06 (Estimated); Last update posted 2011-06-06 (Estimated); Status verified 2010-11

CONDITIONS: Critically Injured Mechanically Ventilated Trauma Patients
Keywords: Trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual method of MHI (Active Comparator)
  Interventions: Other: Usual method of MHI
- Protective MHI (Experimental)
  Interventions: Other: Protective manual hyperinflation

INTERVENTIONS:
Other: Protective manual hyperinflation — Manual hyperinflation for 10 minutes using a Mapleson C circuit and 100% oxygen with volume set at 8mls/kg and positive end expiratory pressure in the circuit appropriate to baseline levels
  Arms: Protective MHI
Other: Usual method of MHI — Manual hyperinflation for 10 minutes using a Mapleson C circuit and 100% oxygen with volume set at 12mls/kg and no positive end expiratory pressure in the circuit
  Arms: Usual method of MHI

SUMMARY:
This single-blinded randomized study aims to compare two methods of manual hyperinflation (protective - moderate tidal volumes with positive end expiratory pressure) and non-protective (large tidal volume and no positive end expiratory pressure) in ventilated acute trauma patients, to investigate the effect on inflammatory markers, lung compliance, oxygenation and sputum volume.

DETAILED DESCRIPTION:
Current evidence in mechanical ventilation supports a "protective lung strategy" that is, smaller tidal volumes and prevention of loss of positive end expiratory pressure (PEEP). There is concern that manual hyperinflation (MHI) may conflict with this strategy and cause volutrauma and atelectrauma potentially leading to biotrauma.

This single-blinded randomized study aims to compare two methods of manual hyperinflation (protective - moderate tidal volumes with positive end expiratory pressure) and non-protective (large tidal volume and no positive end expiratory pressure) in ventilated acute trauma patients, to investigate the effect on inflammatory markers, lung compliance, oxygenation and sputum volume.

ELIGIBILITY:
Inclusion Criteria:

* Trauma patients
* Day 1 of admission to intensive care
* Mechanically ventilated

Exclusion Criteria:

* Pre-existing lung disease
* PEEP > 12.5cmH20
* Nitric oxide in circuit
* Haemodynamically unstable
* Undrained pneumothorax
* Intracranial pressure > 25mmHg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-09; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Interleukin 6 | Change between Baseline and 40 minutes and 70 minutes post baseline
  5 mls of arterial blood will be colected in an EDTA tube, centrifuged and aliquoted within 30 minutes. It will be stored at -80 degrees C and the analysis completed in batches by enzyme linked immunosorbent assay

SECONDARY OUTCOMES:
Tumour necrosis factor alpha | Change from Baseline to 40 minutes and 70 minutes post baseline
  5 mls of arterial blood will be colected in an EDTA tube, centrifuged and aliquoted within 30 minutes. It will be stored at -80 degrees C and the analysis completed in batches by enzyme linked immunosorbent assay
Interleukin 1-beta | Change between baseline and 40 minutes and 70 minutes post baseline
  5 mls of arterial blood will be colected in an EDTA tube, centrifuged and aliquoted within 30 minutes. It will be stored at -80 degrees C and the analysis completed in batches by enzyme linked immunosorbent assay
Interleukin 8 | Change between baseline and 40 minutes and 70 minutes post baseline
  5 mls of arterial blood will be colected in an EDTA tube, centrifuged and aliquoted within 30 minutes. It will be stored at -80 degrees C and the analysis completed in batches by enzyme linked immunosorbent assay
PaO2/FiO2 Oxygenation ratio | Chnge between baseline and 15 minutes and 40 minutes post baseline
  The ratio between the partial pressure of oxygen in arterial blood and the fraction of inspired oxygen which is delivered to the patient.
Static lung compliance | Change between Baseline and 15 minutes and 70 minutes post baseline
  Static lung compliance is the change in volume for any given applied pressure. The formula is Compliance = Change in volume/change in pleural pressure.
  An inspiratory hold will be dialled on the mechanical ventilator and the static lung compliance value will be recorded from the screen.
Mean arterial blood pressure | the change between baseline and every minute during intervention for 10 minutes will be compared
  The mean blood pressure will be recorded from the arterial catheter in situ. This is displayed continuously on the Phillips Intellivue Monitor and will be recorded for the time of intervention
Sputum volume | Immediately at end of intervention
  Sputum will be suctioned at the end of the manual hyperinflation technique by an inline suction catheter using sterile technique into a closed sample jar. This will be weighed on an Acculab Pocket Scale PP401

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Brisbane & Womens Hospital, Brisbane, Queensland, Australia